CLINICAL TRIAL: NCT01548313
Title: The Role of Human Milk in Development of Breast Fed Child's Intestinal Microbiota
Acronym: MYMILK
Status: Completed | Type: Observational
Sponsor: University of Ljubljana (Other)
Collaborators: University Medical Centre Ljubljana (Other)
Responsible Party: Sponsor
Other Study IDs: J4 3606 BF-UL My milk
Record Dates: First submitted 2012-03-05; First posted 2012-03-08 (Estimated); Last update posted 2019-05-01 (Actual); Status verified 2019-04

CONDITIONS: Pregnancy; Lactation
Keywords: human milk; nutrition; breastfed child; microbiota; fatty acids; intestinal microbiota; probiotics
MeSH Terms: conditions — Breast Feeding

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — colostrum, meconium, milk, child's faeces, urine, venous blood
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Pregnant women from Ljubljana region: Women at 3rd trimester of pregnancy living in the Ljubljana region.
- Pregnant women from Izola region: Women at 3rd trimester of pregnancy living in the Izola region.
- Pregnant women from Murska Sobota region: Women at 3rd trimester of pregnancy living in the Murska Sobota region.

SUMMARY:
The ideal food for normal infants is human milk. In addition, breast milk has been shown to be a continuous source of commensal, and⁄or probiotic bacteria to the infant gut where they play a key role in the initiation and development of the gut microbiota. Intestinal colonization is essential for maturation of the gut-associated lymphoid tissue (GALT) and the homeostasis of the intestinal epithelium. Colonization begins immediately after birth, while later the composition of the gut microbiota is affected by feeding practices. Results of some studies suggest that long-chain polyunsaturated fatty acids (LCPUFAs) promote the adhesion of probiotics to mucosal surfaces and along with probiotic bacteria contribute to the regulation of innate and adaptive immune responses and present a link among mother's diet, and microbes. The main purpose of the proposed research is to establish the link among mothers' nutrition, human milk LCPUFAs composition and microbiota and their potential influence on child's gut microbiota development. Pregnant women from three different regions of Slovenia will be involved into the study. Dietary intakes will be assessed during pregnancy, at the beginning of the 3rd trimester of pregnancy, and during lactation, at 4 weeks post partum, by 7-day weighed dietary protocol (7DP). Human milk (colostrum, and mature human milk) and infant's faeces will be sampled twice: at 2 or 3rd day post partum (meconium) and at 4 weeks post partum for the determination of human milk LCPUFAs composition and the assessment of human milk (colostrum und mature) and faeces microbiota. The fatty acid composition of human milk will be analysed by capillary gas-liquid chromatography (GC). Microbiota of milk and faeces will be studied using conventional microbiological and modern molecular approach such as qualitative and quantitative PCR amplification of informative genomic regions, DGGE/TGGE and/or t-RFLP and sequencing. Regular monthly meetings with the researchers will be organised for discussion and advising. Basic health parameters of infants will be followed. Data will be gathered from maternity department medical charts, from regular paediatric health care visits and from especially designed health care diary each mother will keep until the end of her child's first year.

DETAILED DESCRIPTION:
The main goal of the proposed study is to establish the link among mothers' nutrition, human milk LCPUFAs composition and microbiota and their potential influence on child's gut microbiota development. Since the information about the mothers´ diet, about the microbiota and fatty acids composition of human milk, about the faecal microbiota of infants and about the possible mechanisms of eventual transfer of microorganisms from mother to child will be needed to establish these connections. In addition, the influence of vitamine D levels in maternal blood on the bone mineral density in neonates will be determined in the first year of life. The dietary fatty acid composition of plasma lipids in the blood of pregnant women will be assessed.

Mothers and their respective infants will be recruited in the maternity hospitals in three Slovenian regions: Ljubljana, Murska Sobota and Izola. Pregnant women will be invited to participate in the study by informative leaflets during their first visits in the health care centres or gynaecological clinics. All pregnant women who will express interest to participate and fulfilling the participation criteria will be invited to the introductory meeting where they will be informed about the study and will get during 1-hour course, instructions about the writing of 4-day weighed dietary protocol. The meetings will be carried out in the selected regional maternity hospitals. All volunteers willing to participate in the study will get the possibility to get our opinion about their diet during the pregnancy as well as later, during lactation period. The volunteers pregnant women will be also asked to precisely register every probiotic food product or food supplement which they will eat during the last three months of pregnancy and during 4 weeks after delivery.

Informed consent:

The study will be described to pregnant women by principal investigator and/or co-investigators. Following the explanation, the interested pregnant women will be given a written description of the study and the approved informed consent to sign. One copy of the signed document will be provided to the mother and one copy will be retained in the records of the clinical study.

The mothers and respective infants fulfilling the participation criteria for further research will receive written instructions and especially designed health care diary for follow up child's first year health and performance.

The mother will give the second or the third day after the delivery, under the supervision of medical staff, the sample of colostrum. If available, the sample of infant´ meconium will be taken at the same time. Both samples will be subjected to the analyses of microbiota. Samples of mature human milk will be taken under the supervision of medical staff at the first visit of the paediatrician, i.e. 4 weeks after delivery (for determination of fatty acids and microbiota), and again between 12th and 14th week after delivery. Mothers will be asked to bring with also a sample of child's faeces. Cooperation between researchers and respective paediatricians in the health care centres responsible for the infants involved in the study will be also established in order to get insight in the basic data about the development and health of infants.

All infants will be followed up from birth to the age of 12 months according to: a) growth, b) feeding regime, c) development d) bone mineral density and e) health. During their first 12 months of life examinations will take part on six occasions:

* Immediately after birth and during the first three days of life
* At first month (age 28 to 38 days)
* At third month (age 80 to 100 days)
* At sixth month (age 110 to 130 days)
* At ninth month (age 260 to 280 days)
* At twelfth month of age (age 355 to 375 days).

For following growth, development and health standard paediatrics' protocols will be used. Feeding regime will be annotated as:

* exclusively breast feed (BF)
* partially BF (BF + formula)
* only formula. Data will be gathered from maternity department medical charts, from regular paediatric health care visits at the dispensaries and from especially designed health care diary each mother will keep until the end of her child's first year.

The researchers will be responsible for the collecting and keeping records of data about all volunteers involved, of their diaries and of data obtained from paediatricians from health care centres.

Long-chain polyunsaturated fatty acids (LCP), especially docosahexaenoic acid (DHA, C22:6n-3) play an important role for the optimal development and maturation of the nervous system. Adequate supply of LCP, especially of DHA, plays an important role during the period of accelerated growth and differentiation of fetal nervous system during the last trimester of pregnancy and in the first year of life. Recently new Consensus recommendations on dietary fat intake in pregnancy and lactation were issued. We aim to investigate whether dietary intake of Slovenian pregnant and lactating women is in accordance with those new recommendations as well as if their dietary intake is healthy.

Special attention will be given to consumption of LCP and probiotic fermented dairy products. The consumption of probiotic food supplements will be registered as well.

Pregnant women (n=300) from three regions of Slovenia, i.e. Ljubljana with surrounding area (n=100), Izola with surrounding area (n=100) and Murska Sobota with surrounding area (n=100), will be included in the study.

Diet will be examined by the use of 4-day weighed dietary protocol (4DP) which will be done twice:

1. during the pregnancy: in the last third of pregnancy (between 27th and 28th week of pregnancy)
2. during the breast-feeding: 4 weeks after delivery

Objectives:

* to investigate weather nutrition of pregnant and lactating Slovenian women is in accordance with the Central European dietary guidelines
* to investigate whether nutrition of pregnant and lactating Slovenian is in accordance with the recent consensus recommendations on dietary fat intake during pregnancy and lactation
* to evaluate the frequencies of consumption of probiotic products (data will be important for screening the breast milk for the presence of commercially important probiotics)

During the study mothers will continue with their ordinary diet. For all participating women, a lecture and one-hour course with practical examples and demonstrations by the use of a balance and examples of foods, about how to write a 4-day weighed dietary protocol (4DP) will be organised. After the evaluation of diaries, the mothers will also have a possibility to ask for an expert opinion about their diet during the pregnancy as well as during lactation.

At the University Medical Centre of Ljubljana, Division of Paediatrics, the collected data will be evaluated by the help of computer program Prodi 5.2 Expert plus (Stuttgart, Germany). Energy will be expressed as a daily intake in kcal and MJ. Nutrient intakes will be expressed in (micro) grams/day, while carbohydrate, protein and fat intakes will also be expressed as a percentage of contribution to the daily energy intake. The intake of sea fish and the fatty acids, especially of DHA as well as the intake of probiotic products will be also precisely evaluated.

The nutrition of pregnant and breast-feeding mothers will be compared with the Central European reference intakes, D-A-CH (D-German, A-Austrian; CH-Swiss) Reference Values for Nutrient Intake which are official in Slovenia since 2004. The intake of fats, especially of DHA, will be compared with the recent consensus recommendations on fat intake during pregnancy and lactation. As the D-A-CH Reference Values do not define the maximum amount of daily sodium and sugar intake, we will compare the sodium and sugar intake with the joint WHO/FAO recommendations (population nutrient intake goal for sodium: < 2 g/day and for free sugars: < 10 % of daily energy intake). The proportion of n-3 LCP in plasma lipids of pregnant women will be compared to their diet. The blood obtained from the pregnant women will be analysed for the content of D vitamine and fatty acids composition of plasma lipids. The purpose of these additional test will be

* to establish whether the consumption of marine fish as well as supplements containing fish oil or unicellular organisms with n-3 LCP (EPA and DHA) (capsules, syrups), before and during pregnancy affects the increase of n-3 LCP in plasma lipids, and
* to assess the influence of dietary factors on bone mineral density in women, and the influence of the levels of vitamin D in the blood of mothers to the bone mineral density in neonates.

Among pregnant women included in the study of diet of pregnant and breast-feeding mothers in Slovenia, 40 mothers from each of regions will be randomly selected, after evaluating of inclusion and exclusion criteria, for the investigation of fatty-acid composition and microbial composition of human milk as well as analysis of faecal microbiota of infants.

Objectives:

* the assessment of fatty acids composition of human milk, with emphasis on LCPUFAs
* the investigation of the correlation between dietary DHA intake (4DP) and its content (wt. %) in mature human milk
* the assessment of microbial diversity of human colostrum and milk microbiota, with emphasis on bifidobacteria and lactic acid bacteria - potential probiotics
* the assessment of the prevalence of bacteriocin producing lactic acid bacteria in the natural microbiota of human colostrum and milk
* the assessment of microbial diversity of child's meconium and faeces
* comparison of milk and child's faecal microbiota

Statistic evaluation of final results will be performed by independent statistician from the Institute of Biostatistics and Medical informatics which has been already included in the preparation of the protocols of clinical studies (WP1).

ELIGIBILITY:
Inclusion Criteria:

* healthy pregnant women
* living in Slovenia
* intend to fully breast-feed their babies at least 6 weeks after delivery
* willing to write a 4-day weighted dietary protocol (7DP) twice: during pregnancy and again at 4 weeks post partum

Exclusion Criteria:

* autoimmune chronic diseases
* acute and chronic infections
* increased risk for premature delivery

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Slovenian, otherwise healthy pregnant women, plan to fully breastfeed their baby for at least 6 weeks, willingness to write a 7-day weighted dietary protocol (7DP) twice: during pregnancy and again at 4 weeks post partum.
Sampling Method: Probability Sample
Enrollment: 294 (Actual)
Dates: Start 2010-05; Primary Completion 2013-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Effect of nutrition patterns of pregnant and lactating women on fatty acid composition of milk and plasma lipids, vitemine D in blood, bone density and composition of microbiota of colostrum, milk, meconium and child's faeces | from 27th-28th week of pregnancy to 12th-14th week post partum
  Nutrition patterns of pregnant and lactating women will be assessed by 4-day weighed dietary protocol (27.-28. week of pregnancy and 4 weeks after delivery). Fatty acids composition of milk, will be determined 4 weeks post partum and between 12th and 14th week post partum. Microbial composition of human colostrum, milk, child's meconium and faeces with emphasis on bifidobacteria and lactic acid bacteria will be determined 2nd- 3rd day post partum, at 4 weeks post partum and 12th-14th week post partum). The vitamin D and fatty acids in blood will be determined at 27th-37th week of pregnancy.

SECONDARY OUTCOMES:
Health and development of a child | The first 12 months post partum
  Growth, type of nutrition, development and health status will be observed. The babies will be examined six times: at birth, at 1st month (between 28th and 38th day), at 3rd month (between 80th and 100th day), at 6th month (between 110th and 130th day), at 9th month (between 260th and 280th day) and at 12th month (between 355th and 375th day).The bone density will be determined at birth and at 1st, 3rd and 12th months.

CONTACTS AND LOCATIONS:
Overall Officials: Irena Rogelj, Prof., Principal Investigator — University of Ljubljana
Locations (1):
- University Medical Centre Ljubljana, Division of Paediatrics, Department of Neonatology, Ljubljana, Slovenia

IPD SHARING:
Plan to Share IPD: No
Scientific articles

REFERENCES:
- [Result] Obermajer T, Grabnar I, Benedik E, Tusar T, Robic Pikel T, Fidler Mis N, Bogovic Matijasic B, Rogelj I. Microbes in Infant Gut Development: Placing Abundance Within Environmental, Clinical and Growth Parameters. Sci Rep. 2017 Sep 11;7(1):11230. doi: 10.1038/s41598-017-10244-x. PMID 28894126
- [Result] Obermajer T, Lipoglavsek L, Tompa G, Treven P, Lorbeg PM, Matijasic BB, Rogelj I. Correction: Colostrum of Healthy Slovenian Mothers: Microbiota Composition and Bacteriocin Gene Prevalence. PLoS One. 2015 Jun 29;10(6):e0132201. doi: 10.1371/journal.pone.0132201. eCollection 2015. No abstract available. PMID 26120836
- [Result] Soltirovska Salamon A, Benedik E, Bratanic B, Velkavrh M, Rogelj I, Fidler Mis N, Bogovic Matijasic B, Paro-Panjan D. Vitamin D Status and Its Determinants in Healthy Slovenian Pregnant Women. Ann Nutr Metab. 2015;67(2):96-103. doi: 10.1159/000439093. Epub 2015 Sep 5. PMID 26340437
- [Result] Benedik E, Korousic Seljak B, Hribar M, Rogelj I, Bratanic B, Orel R, Fidler Mis N. Comparison of a Web-Based Dietary Assessment Tool with Software for the Evaluation of Dietary Records. Zdr Varst. 2015 Mar 13;54(2):91-7. doi: 10.1515/sjph-2015-0014. eCollection 2015 Jun. PMID 27646914
- [Result] Benedik E, Korousic Seljak B, Simcic M, Rogelj I, Bratanic B, Ding EL, Orel R, Fidler Mis N. Comparison of paper- and web-based dietary records: a pilot study. Ann Nutr Metab. 2014;64(2):156-66. doi: 10.1159/000363336. Epub 2014 Aug 9. PMID 25116257
- [Result] Robic T, Benedik E, Fidler Mis N, Bratanic B, Rogelj I, Golja P. Challenges in determining body fat in pregnant women. Ann Nutr Metab. 2013;63(4):341-9. doi: 10.1159/000358339. Epub 2014 Mar 6. PMID 24603563
- [Result] Obermajer T, Pogacic T. Commentary: Relationship between Milk Microbiota, Bacterial Load, Macronutrients, and Human Cells during Lactation. Front Microbiol. 2016 Aug 17;7:1281. doi: 10.3389/fmicb.2016.01281. eCollection 2016. No abstract available. PMID 27581429